CLINICAL TRIAL: NCT04882735
Title: A Phase 3, Open-Label, Multicenter, Single-Arm Study to Evaluate the Efficacy and Safety of Acoramidis in Subjects with Symptomatic Transthyretin Amyloid Polyneuropathy (ATTRibute-PN Study)
Brief Title: Efficacy and Safety of Acoramidis (AG10) in Subjects with Transthyretin Amyloid Polyneurophathy (ATTRibute-PN)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision to cancel study
Sponsor: Eidos Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG10-334
Record Dates: First submitted 2021-04-29; First posted 2021-05-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-01

CONDITIONS: Transthyretin-Related (ATTR) Familial Amyloid Polyneuropathy
Keywords: TTR; ATTR-PN; Familial ATTR-PN; Amyloidosis; Amyloid; Transthyretin; Polyneuropathy; TTR-mediated amyloidosis; Amyloidosis, hereditary; Familial Amyloid Polyneuropathies; Amyloidosis, Hereditary, Transthyretin-Related
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis; Alzheimer Disease; Polyneuropathies; Amyloidosis, Familial; Amyloidosis, Hereditary, Transthyretin-Related | interventions — attruby

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Acoramidis HCI 800 mg (two 400mg tablets) (Experimental): TTR stabilizer administered orally twice daily (BID)
  Interventions: Drug: Acoramidis

INTERVENTIONS:
Drug: Acoramidis — TTR stabilizer administered orally twice daily (BID)
  Other Names: AG10

SUMMARY:
Phase 3 efficacy and safety of acoramidis in subjects with symptomatic Transthyretin Amyloid Polyneuropathy (ATTR-PN)

DETAILED DESCRIPTION:
Transthyretin amyloid polyneuropathy (ATTR-PN), also called "Familial Transthyretin-Mediated Amyloid Polyneuropathy (FAP)" is a hereditary condition caused by mutations in the TTR gene. It is estimated that around 10,000 people in the world are affected.

In ATTR-PN, amyloid builds up in the nerves that detect temperature, pain, and touch. Patients with ATTR-PN can experience a loss of sensation, tingling, numbness, or pain in the hands and feet (also called peripheral neuropathy).

In this study Eidos, a BridgeBio Company, is researching the investigational drug acoramidis (AG10) hydrochloride (HCl) 800mg administered orally twice a day. Through the study, Eidos/BridgeBio wants to evaluate the efficacy and safety of acoramidis in patients with ATTR-PN.

The primary outcome of the study is to determine the efficacy of acoramidis in the treatment of subjects with symptomatic transthyretin amyloid polyneuropathy (ATTR-PN).

At the end of 18 months, participants will be eligible to continue to receive acoramidis to evaluate the long-term safety and tolerability of acoramidis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 to ≤90 years of age;
* Have Stage I or II symptoms (polyneuropathy disability [PND] ≤IIIb) of ATTR-PN and an established diagnosis of ATTR-PN as defined by physical examination findings and/or neurophysiological test findings consistent with the diagnosis of ATTR-PN;
* Have an NIS of 5 to 130 (inclusive) during Screening;
* Have a nerve conduction studies (NCS) score (sum of the sural sensory nerve action potential [SNAP], tibial compound muscle action potential (CMAP), ulnar SNAP, ulnar CMAP, and peroneal CMAP) of ≥2 points during Screening. NCS is a component of mNIS+7;
* Have a mutation consistent with ATTR-PN either documented in medical history or confirmed by genotyping obtained at Screening prior to enrollment. No genetic testing is needed for subjects who are recipients of domino liver transplants;
* Have an anticipated survival of >2 years in the opinion of the investigator;
* Have Karnofsky performance status ≥60 %.

Exclusion Criteria:

* Had a prior liver transplantation or is planning to undergo liver transplantation with a wild-type organ graft as treatment for symptomatic ATTR-PN during the study period. Note: Recipients of a "domino" liver transplant from an ATTR-PN donor who have developed ATTR-PN mediated by their graft are allowed under this protocol, as long as re-transplantation to treat ATTR-PN is not planned during the study period and meets all other eligibility criteria;
* Has sensorimotor or autonomic neuropathy not related to ATTR-PN; for example, due to autoimmune disease or monoclonal gammopathy, malignancy, or alcohol abuse;
* Has Vitamin B-12 levels below the lower limit of normal (LLN) at Screening;
* Has clinical evidence of untreated hyperthyroidism or hypothyroidism;
* Has leptomeningeal TTR amyloidosis;
* Has Type 1 diabetes;
* Has had Type 2 diabetes for ≥5 years;
* Has a documented case of hepatitis B or C at Screening;
* Known history of human immunodeficiency virus (HIV) infection;
* Has NYHA heart failure classification >Class II;
* Had acute coronary syndrome, uncontrolled cardiac arrhythmia, or a stroke within 90 days prior to Screening;
* Has estimated glomerular filtration rate (eGFR) by Modification of Diet for Renal Disease (MDRD) formula <30 mL/min/1.73 m2 at Screening;
* Has abnormal liver function tests at Screening, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × upper limit of normal (ULN) or total bilirubin >3 × ULN;
* Had a malignancy within 2 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated;
* Has known hypersensitivity to acoramidis, its metabolites, or formulation excipients.
* Is currently undergoing treatment for ATTR-PN with tafamidis, or patisiran, inotersen, or other knockdown agents, marketed drug products lacking a labeled indication for ATTR-PN (e.g., diflunisal, doxycycline), natural products or derivatives used as unproven therapies for ATTR-PN (e.g., green tea extract ,tauroursodeoxycholic acid [TUDCA]/ursodiol), within 14 days, or 14 days for tafamidis or 90days for patisiran and 180 days for inotersen prior to dosing.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Month 18 in mNIS+7 | 18 Months
  To determine the efficacy of acoramidis in subjects with symptomatic transthyretin amyloid polyneuropathy (ATTR-PN) by evaluating the change in Modified Neuropathy Impairment Score +7 (mNIS+7) from baseline to 18 months.
Safety: TESAEs will be used to evaluate the long-term safety and tolerability of acoramidis administered to subjects with symptomatic polyneuropathy (ATTR-PN) | 60 Months
  To evaluate the long-term safety and tolerability of acoramidis administered to subjects with symptomatic transthyretin amyloid polyneuropathy (ATTR-PN)
Safety: Adverse Events leading to treatment discontinuation will be used to evaluate the long-term safety and tolerability of acoramidis administered to subjects with symptomatic polyneuropathy (ATTR-PN) | 60 Months
  To evaluate the long-term safety and tolerability of acoramidis administered to subjects with symptomatic transthyretin amyloid polyneuropathy (ATTR-PN)
Safety: Adverse Events will be used to evaluate the long-term safety and tolerability of acoramidis administered to subjects with symptomatic polyneuropathy (ATTR-PN) | 60 Months
  To evaluate the long-term safety and tolerability of acoramidis administered to subjects with symptomatic transthyretin amyloid polyneuropathy (ATTR-PN)
Safety: Incidence of abnormal physical exam will be used to evaluate the long-term safety and tolerability of acoramidis administered to subjects with symptomatic polyneuropathy (ATTR-PN) | 60 Months
  To evaluate the long-term safety and tolerability of acoramidis administered to subjects with symptomatic transthyretin amyloid polyneuropathy (ATTR-PN)
Safety: Incidence of abnormal vital signs will be used to evaluate the long-term safety and tolerability of acoramidis administered to subjects with symptomatic polyneuropathy (ATTR-PN) | 60 Months
  To evaluate the long-term safety and tolerability of acoramidis administered to subjects with symptomatic transthyretin amyloid polyneuropathy (ATTR-PN)
Safety: Columbia-Suicide Severity Rating Scale (C-SSRS) will be used to evaluate the long-term safety and tolerability of acoramidis administered to subjects with symptomatic polyneuropathy (ATTR-PN) | 60 Months
  To evaluate the long-term safety and tolerability of acoramidis administered to subjects with symptomatic transthyretin amyloid polyneuropathy (ATTR-PN)

SECONDARY OUTCOMES:
Change from baseline to Month 18 in Norfolk QOL-DN | 18 Months
  To evaluate the effects of acoramidis in subjects with symptomatic ATTR-PN on Norfolk Quality of Life Questionnaire-Diabetic Neuropathy (Norfolk QOL-DN)
Change from baseline to Month 18 in mBMI | 18 Months
  To evaluate the effects of acoramidis in subjects with symptomatic ATTR-PN on Modified body mass index (mBMI)
Change from baseline to Month 18 in COMPASS-31 | 18 Months
  To evaluate the effects of acoramidis in subjects with symptomatic ATTR-PN on Composite Autonomic Score (COMPASS-31)

CONTACTS AND LOCATIONS:
Overall Officials: Mark McGovern, RN, CCRN, Study Director — Eidos Therapeutics, a BridgeBio company

IPD SHARING:
Plan to Share IPD: No